CLINICAL TRIAL: NCT06155461
Title: Preoperative Ultrasonographic Evaluation of Caval Aorta Diameter Index as a New Predictor for Hypotension After Induction of General Anesthesia in Geriatric Patients
Brief Title: Preoperative Ultrasonographic Evaluation of Caval Aorta Diameter Index
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Other Study IDs: Anaesth._0319/2023Med.Research
Record Dates: First submitted 2023-11-19; First posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Hypotension; Geriatric Patients; Anesthesia
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Preoperative Ultrasonographic Evaluation of Caval Aorta Diameter Index — to evaluate the ability of preoperative ultrasound measurements of IVC to aorta diameter index and the inferior vena cava collapsibility index (IVCCI) for predicting post induction hypotension after general anesthesia in geriatric patients.

SUMMARY:
General anesthesia is frequently used in daily clinical practice. Elderly patients often require a higher level of care than younger patients during the perioperative period, with higher health care costs.

Strategies to optimize anesthesia care to reduce complications and improve outcomes in elderly surgical patients will also be of great value to the individual patients and society.

DETAILED DESCRIPTION:
Prevention of an undesired hypotensive event has a key role in providing patient safety. Patients' susceptibility to intra-operative hypotension can be influenced by the pre-operative volume status.

Despite worldwide improvement in preoperative optimization and changing practices, promoting the avoidance of unnecessary fasting and mechanical bowel preparation, optimized fluid therapy remains the cornerstone of treatment with excellent effectiveness.

The earlier, non-invasive and bedside investigation for assessment of volume status will enhance the effective prevention and management of post-induction hypotension and hence better clinical outcome .

Several methodologies have been tried with a specific goal to predict post-induction hypotension, including heart rate variability (HRV), passive leg raise test and perfusion index.

Despite this, assessing intravascular volume status is still challenging matter. Therefore, the aim of this study will be to compare between the collapsibility index of the inferior vena cava (IVCCI) and IVC to aorta diameter index (IVCD: AoD index) as a potential screening tool to identify patients who are vulnerable to hypotensive events related to general anesthesia.

IVCCI has been tested before in several studies as a predictor of post-induction hypotension. However, IVCD: AoD index has not been investigated before for prediction of hypotension after induction of general anesthesia in elderly. Among the earliest studies to assess the IVCD: AoD index was carried out by Kodiak et al., in hypovolemic patients.

Additionally, it has been investigated for predicting the postspinal anesthesia hypotension and showed promising results

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ( 60 - 85 ) years old of both sexes with American Society of Anesthesiologists (ASA) physical status I-II and scheduled for elective surgeries under general anesthesia.

Exclusion Criteria:

1. Refusal to join the study.
2. Mental and psychiatric disorders (un co-operative patients).
3. Emergency operations
4. ASA physical status > II
5. Dyspnea, respiratory distress, un-compensated respiratory disease (generalized wheezes, defective functional capacity, peripheral O2 saturation less than 90% on room air )
6. patients with uncontrolled hypertension, Systolic blood pressure ≥ 180 mmHg
7. IVC non visualized
8. Patients with increased intra-abdominal pressure (intra-abdominal mass compressing IVC).
9. anticipated or accidental discovered difficult airway
10. patients taking angiotensin converting enzyme inhibitors or angiotensin receptors blockers, documented heart failure, elevated pulmonary arterial pressure > 40 mmHg, significant valvular heart disease, significant carotid stenosis, peripheral vascular diseases, unstable angina or cardiac ejection fraction less than 40%, implanted pacemaker or cardioversion , known cases of abdominal aortic abnormality as aneurysm or previous operations.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective surgery under general anesthesia, ASA I, II
Sampling Method: Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-15 (Estimated)

PRIMARY OUTCOMES:
Evaluate the predictive value of pre-induction IVC | 5 minutes
  Area under receiver operating characteristic curves (AUROC) of the preoperative IVCCI inprediction of post-induction hypotension

SECONDARY OUTCOMES:
Incidence of post-induction hypotension | 5 minutes
  Correlation between each of maximum aortic diameter with the percentage of the maximum decrease in mean arterial pressure after induction of anesthesia
Correlation between each of IVC collapsibility index with the percentage of the maximum decrease in mean arterial pressure after induction of anesthesia | 5 minutes
  Correlation between each of IVC collapsibility index with the percentage of themaximum decrease in mean arterial pressure after induction of anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Saied, Professor, Study Chair — Al-Azhar University, Faculty of medicine for boys
Locations (1):
- Al-Azhar University hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided